CLINICAL TRIAL: NCT04230369
Title: Internet-delivered Cognitive Behaviour Therapy for Anxiety Related to Asthma: A Randomized Controlled Trial
Brief Title: Internet-delivered CBT for Anxiety Related to Asthma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Catarina Almqvist Malmros, Professor, MD, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MANTRA03
Record Dates: First submitted 2019-12-20; First posted 2020-01-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Asthma; Anxiety
MeSH Terms: conditions — Asthma; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The participants will be randomised to immediate internet-CBT or 4 months of treatment as usual before cross-over to internet-CBT.
Who Masked: Outcomes Assessor
Masking Description: All assessments will be conducted by participants over the internet, why there can be no influence from study staff during data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-CBT (Experimental): The internet-CBT will comprise 8 weekly modules with therapist-support, encouraging exposure for fear of asthma symptoms while ensuring a stable asthma medication through a written medical plan on medical adherence Participants work independently from home with the treatment and receive weekly support from their psychologist through written messages online.
  Interventions: Behavioral: Exposure-based Internet-CBT
- Treatment as usual (Other): Patients randomized to treatment as usual will receive the same medical information that participants in the Internet-CBT get, with physiological information about asthma and the importance of medical adherence to achieve well controlled asthma, but without the exposure-based treatment and no therapist support. All participants in both conditions can use any other available treatment, but psychological, from pre-assessments to 2 months after treatment completion. Participants in this arm will be crossed over to Internet-CBT after the primary endpoint at to 2 months follow up.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Exposure-based Internet-CBT — Internet-CBT for anxiety-related asthma 8 weekly modules of CBT delivered over the internet and targeting enhanced function and decreased symptoms of anxiety. Participants work independently from home with the treatment and receive support from experienced Internet-CBT Psychologists through written messages in the secure platform. All participants in both conditions can use any other available treatment (TAU), but psychological, from pre-assessments to 2 months after treatment completion.
  Other Names: Online exposure therapy
  Arms: Internet-CBT
Other: Treatment as usual — Patients randomized to treatment as usual will receive the same medical information that participants in the Internet-CBT get, with physiological information about asthma and the importance of medical adherence to achieve well controlled asthma, but without the exposure-based treatment and no therapist support. All participants in both conditions can use any other available treatment (TAU), but psychological, from pre-assessments to 2 months after treatment completion.
  Other Names: TAU
  Arms: Treatment as usual

SUMMARY:
This is a randomized controlled trial to investigate efficacy of a internet-delivered CBT for anxiety related to asthma.

DETAILED DESCRIPTION:
Asthma is one of the most common chronic diseases and is often associated with anxiety. In a two prior studies (ClinicalTrials.gov ID: NCT03158194; NCT03486756) a protocol for exposure-based cognitive behaviour therapy (CBT) for anxiety related to asthma was developed, and standardised to an internet-delivered format and tested for feasibility and acceptability as an internet-CBT. The aim of the current study is to evaluate the efficacy of exposure-based Internet-CBT for anxiety related to asthma compared to Treatment as Usual (TAU). The plan is to include 90 participants consecutively during 2020.

ELIGIBILITY:
Inclusion Criteria:

* asthma diagnosed by a physician
* worry about asthma or limitations in daily life due to asthma at

Exclusion Criteria:

* a serious psychiatric condition; e.g., suicidality, psychosis or severe substance addiction
* chronic obstructive pulmonary disease (COPD) or other chronic airway disorders other than asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Catastrophizing about asthma Scale | Time Frame: Baseline to 16 weeks; baseline to 36 weeks; baseline to 12 months.
  Change in catastrophizing cognitions about asthma measured with a self-rating scale at baseline, weekly during treatment, at 16 weeks, 36 weeks and 12 months for analysis of effect.

SECONDARY OUTCOMES:
Asthma control test | Time Frame: Baseline to 16 weeks; baseline to 36 weeks; baseline to 12 months.
  Change in asthma control measured with a self-rating scale at baseline, weekly during treatment, at 16 weeks, 36 weeks and 12 months for analysis of effect.
Penn State Worry Questionnaire | Time Frame: Baseline to 8 weeks; baseline to 16 weeks; baseline to 36 weeks; baseline to 12 months.
  Change in subjective worry measured with a self-rating scale measured with a self-rating scale at baseline, at 16 weeks, 36 weeks and 12 months for analysis of effect.
Asthma Quality of Life Questionnaire | Time Frame: Baseline to 8 weeks; baseline to 16 weeks; baseline to 36 weeks; baseline to 12 months.
  Change in asthma-related quality of life measured with a self-rating scale at baseline, at 16 weeks, 36 weeks and 12 months for analysis of effect.
Short Health Anxiety Inventory (SHAI) | Time Frame: Baseline to 8 weeks; baseline to 16 weeks; baseline to 36 weeks; baseline to 12 months.
  Change in health anxiety measured with a self-rating scale at baseline, at 16 weeks, 36 weeks and 12 months for analysis of effect.
Perceived Stress Scale | Time Frame: Baseline to 16 weeks; baseline to 36 weeks; baseline to 12 months.
  Change in perceived stress measured with a self-rating scale at baseline, weekly during treatment, at 16 weeks, 36 weeks and 12 months for analysis of effect.
Fear of Asthma Symptoms | Time Frame: Baseline to 16 weeks; baseline to 36 weeks; baseline to 12 months.
  Change in fear of asthma symptoms measured with a self-rating scale at baseline, weekly during treatment, at 16 weeks, 36 weeks and 12 months for analysis of effect.
Asthma Behaviour Checklist | Time Frame: Baseline to 16 weeks; baseline to 36 weeks; baseline to 12 months.
  Change in behaviour related to asthma anxiety measured with a self-rating scale at baseline, weekly during treatment, at 16 weeks, 36 weeks and 12 months for analysis of effect.
Insomnia Severity Index | Time Frame: Baseline to 16 weeks; baseline to 36 weeks; baseline to 12 months.
  Change in insomnia measured with a self-rating scale at baseline, at 16 weeks, 36 weeks and 12 months for analysis of effect.
Patient Health Questionnaire-9 | Time Frame: Baseline to 8 weeks; baseline to16 weeks; baseline to 36 weeks; baseline to 12 months.
  Change in depression measured with a self-rating scale at baseline, at 16 weeks, 36 weeks and 12 months for analysis of effect.
WHODAS | Time Frame: Baseline to 8 weeks; Baseline to 16 weeks; baseline to 36 weeks; baseline to 12 months.
  Change in health related quality of life for health economic evaluation measured with a self-rating scale at baseline, at 16 weeks, 36 weeks and 12 months for analysis of effect.
Brunnsviken quality of life scale | Time Frame: Baseline to 8 weeks; baseline to16 weeks; baseline to 36 weeks; baseline to 12 months.
  Change in general quality of life measured with a self-rating scale at baseline, at 16 weeks, 36 weeks and 12 months for analysis of effect.
Treatment Inventory of Costs in Patients | Time Frame: Baseline to 8 weeks; baseline to16 weeks; baseline to 36 weeks; baseline to 12 months.
  Change in health consumption measured with a self-rating scale at baseline, postreatment and at 16 weeks for analysis of effect.
Asthma Tuner | Time Frame: Baseline to 8 weeks; baseline to16 weeks.
  Change in FEV1 measured with a digital spirometer at baseline, posttreatment and at 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Catarina A Almqvist, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of Medical Epidemiology and Biostatistics, Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bonnert M, Nash S, Andersson EM, Bergstrom SEE, Gorling J 1, Janson C, Sarnholm J, Almqvist C. Online cognitive behaviour therapy for asthma-related anxiety: a randomised controlled trial. Thorax. 2026 Jan 6:thorax-2025-223886. doi: 10.1136/thorax-2025-223886. Online ahead of print. PMID 41494908
- [Derived] Bonnert M, Nash S, Andersson EM, Bergstrom SE, Janson C, Almqvist C. Internet-delivered cognitive-behaviour therapy for anxiety related to asthma: study protocol for a randomised controlled trial. BMJ Open Respir Res. 2024 May 27;11(1):e002035. doi: 10.1136/bmjresp-2023-002035. PMID 38802281